CLINICAL TRIAL: NCT02300350
Title: A Phase 1, Single-center, Open-label, Two-period, Single-sequence, Drug-drug Interaction Study to Evaluate the Effects of Multiple-dose LX4211 on the Pharmacokinetics of Single-dose Digoxin (Lanoxin®), a Sensitive P-glycoprotein (P-gp) Substrate, in Healthy Male and Female Subjects
Brief Title: DDI Study With Multiple-dose LX4211 and Single Dose Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-114-NRM; LX4211.114 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 0.5 mg single-dose oral digoxin administration
  Interventions: Drug: Treatment A digoxin
- Treatment B (Experimental): 400 mg oral LX4211 qd administration
  Interventions: Drug: Treatment B LX4211
- Treatment C (Experimental): 0.5 mg single-dose oral digoxin administration + 400 mg oral LX4211 qd administration
  Interventions: Drug: Treatment C Digoxin + 400 mg LX4211 administered concomitantly

INTERVENTIONS:
Drug: Treatment A digoxin — 0.5 mg digoxin administered on Day 1 and Day 20
  Arms: Treatment A
Drug: Treatment B LX4211 — 400 mg LX4211 administered daily on Day 14 through Day 25
  Arms: Treatment B
Drug: Treatment C Digoxin + 400 mg LX4211 administered concomitantly — 0.5 mg Digoxin + 400 mg LX4211 administered concomitantly on Day 20
  Arms: Treatment C

SUMMARY:
This study will be conducted as a single-center, open-label, 2-period, single-sequence, drug-drug interaction study to assess the effects of multiple dose LX4211 (400 mg administered as 2 × 200-mg tablets qd × 12 days) on the PK of single-dose digoxin (2 × 0.25-mg tablets) in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 to ≤55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mmHg; diastolic blood pressure, 50-90 mmHg; heart rate, 45-100 bpm
* Body mass index (BMI) ≥18 and ≤32 kg/sq m
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings that, in the opinion of the Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results
* History of clinically significant arrhythmias
* History of cardiac arrhythmias or palpitations associated with presyncope, syncope, or a family history of sudden cardiac death
* Use of any medications or supplements/supratherapeutic doses of vitamins within 14 days prior to the first dose administration and throughout the duration of the study
* Receipt of any investigational agent or study drug within 30 days prior to Screening
* Receipt of any protein- or antibody-based therapeutic agents within 3 months prior to Screening
* Prior exposure to LX4211
* Use of tobacco, smoking cessation products, or products containing nicotine within 3 months prior to Screening and for the duration of the study
* History of any serious adverse reaction or hypersensitivity to any inactive component of LX4211 or digoxin
* Existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism, or excretion of LX4211 or digoxin
* History of any major surgery within 6 months or anticipated surgery prior to Day 1
* History of any clinically significant hypoglycemia or hyperglycemia
* History of renal disease, or significantly abnormal kidney function test at Screening
* History of hepatic disease, or significantly abnormal liver function tests at Screening
* History of any clinically relevant psychiatric, renal, hepatic, pancreatic, endocrine, cardiovascular, neurological, hematological, or GI abnormality
* History of any active infection within 14 days prior to Day 1
* History of alcohol or substance abuse within 2 years prior to Screening
* Positive hepatitis panel
* Donation or loss of >500 mL of blood or blood product within 3 months prior to Screening
* Women who are breastfeeding or are planning to become pregnant during the study, or women who have a positive serum pregnancy test
* Positive urine glucose at Screening
* Positive urine screen for drugs of abuse and cotinine at Screening, Day -1, or Day 13
* Inability or difficulty swallowing whole tablets
* Unable or unwilling to cooperate with the Investigator for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC | Day 1-Day 7, Day 20-26

SECONDARY OUTCOMES:
Adverse Events | Day 1-Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Dallas, Texas, United States